CLINICAL TRIAL: NCT05471804
Title: Psychological Effects of 8 Weeks Supplementation With Sceletium Tortuosum Extract (Zembrin™): a Randomised, Double Blind, Placebo-controlled, Parallel-groups Trial
Brief Title: Psychological Effects of 8 Weeks Supplementation With Sceletium Tortuosum Extract
Acronym: ZEMBRIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northumbria University (Other)
Collaborators: HG&H Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Emma Wightman, Associate Professor, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 61CC1
Record Dates: First submitted 2022-07-13; First posted 2022-07-25 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Cognitive Change; Stress, Psychological
Keywords: Zembrin; Sceletium tortuosum; COMPASS
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo control (Placebo Comparator): An inert tablet with the same physical appearance as the experimental intervention tablet
  Interventions: Dietary Supplement: Sceletium tortuosum
- Zembrin (Experimental): 25 mg per day of Sceletium tortuosum extract (Zembrin®)
  Interventions: Dietary Supplement: Sceletium tortuosum

INTERVENTIONS:
Dietary Supplement: Sceletium tortuosum — Zembrin® is a proprietary low-alkaloid extract of Sceletium tortuosum, often consumed by healthy humans in order to decrease anxiety and stress and improve cognitive function under stressful situations
  Other Names: Zembrin

SUMMARY:
This study employs a randomized controlled trial to test the cognitive enhancing and stress relieving potential of the product Zembrin® in healthy adults when consumed over an 8 week period.

DETAILED DESCRIPTION:
The aim of the proposed randomized, double-blind, placebo-controlled, parallel groups study is to assess the effects of 8 weeks supplementation with Zembrin®, in 30-50 year old healthy adults, on cognitive function, mood, psychological and physiological stress responses during a laboratory stressor, fatigue and sleep quality. The trial will utilize the COMPASS cognitive assessment system and a range of mood measures and will employ the Observed Multitasking Stressor (OMS), with psychological state and physiological responses assessed before and after, and cognitive function assessed during, the stressor. The cognitive/mood assessments will take place prior to (Day -1 with respect to treatment) and after 8 weeks supplementation with Zembrin. An interim mood/fatigue assessment will take place online (Cognimapp) with a baseline measurement collected between the screening visit and Day -1 and post dose measurements collected after 7 and 28 days 1 and 4 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must self-assess themselves as being in good health Aged 30 to 50 years at the time of giving consent

Exclusion Criteria:

Participants are not eligible to take part if they:

* Have any pre-existing medical condition/illness which will impact taking part in the study NOTE: the explicit exceptions to this are controlled hay fever, high cholesterol and reflux-related conditions. There may be other, unforeseen, exceptions and these will be considered on a case-by-case basis; i.e. participants may be allowed to progress to screening if they have a condition/illness which would not interact with the active treatments or impede performance.
* Are currently taking prescription medications NOTE: the explicit exceptions to this are contraceptive treatments for female participants, those medications used in the treatment of reflux-related conditions; and those taken 'as needed' in the treatment of asthma and hay fever. As above, there may be other instances of medication use which, where no interaction with the active treatments is likely, and which would not be expected to have any impact on brain function, participants may be able to progress to screening.
* Have high blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Have a Body Mass Index (BMI) outside of the range 18.5-35 kg/m2
* Are pregnant, seeking to become pregnant or lactating.
* Are menopausal/post-menopausal
* Have learning and/or behavioural difficulties such as dyslexia or ADHD
* Have a visual impairment that cannot be corrected with glasses or contact lenses (including colour-blindness)
* Smoke tobacco or vape nicotine or use nicotine replacement products
* Take any illicit social drugs, including cannabis
* Have excessive caffeine intake (>500 mg per day)
* Have relevant food intolerances/ sensitivities
* Have taken antibiotics within the past 4 weeks
* Have taken dietary supplements eg. Vitamins, omega 3 fish oils, herbal extracts, cannabadiol etc. in the last 4 weeks (Note: participation is possible following a 4 week supplement washout prior to participating and for the duration of the study on the proviso that the supplements they are taken are out of choice and not medically prescribed or advised). Existing and consistent use of vitamin D supplements and protein shakes are permitted
* Have any health condition that would prevent fulfilment of the study requirements (this includes non-diagnosed conditions for which no medication may be taken)
* Are unable to complete all of the study assessments
* Are currently participating in other clinical or nutrition intervention studies, or have in the past 4 weeks
* Has been diagnosed with/ undergoing treatment for alcohol or drug abuse in the last 12 months
* Have been diagnosed with/ undergoing treatment for a psychiatric disorder in the last 12 months
* Suffers from frequent migraines that require medication (more than or equal to 1 per month)
* Sleep disorders or are taking sleep aid medication
* Any known active infections
* Have oral disease
* Does not have a bank account (required for payment)
* Are non-compliant with regards treatment consumption

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Subjective stress | 56 days
  This outcome will be assessed via changes on the Perceived Stress Scale (PSS). This is a 10 item scale scored from 0 (NEVER) to 4 (very often) with a higher score indicating greater stress.

SECONDARY OUTCOMES:
Mental fatigue | 56 days
  This outcome will be assessed via changes on the Multidimensional Fatigue Inventory (MFI-20). This is a 20 item questionnaire scored from 1 (yes, that is true) to 7 (no, that is not true) with higher scores indicating more fatigue.
Subjective happiness | 56 days
  This outcome will be assessed via changes on the Oxford Happiness Questionnaire (OHQ). This is a 29 item questionnaire scored from 1 (strongly disagree) to 6 (strongly agree) with a higher score indicating greater happiness.
Subjective alertness | 56 days
  This outcome will be assessed via changes on the Visual Analogue Scale (VAS) for alertness. This VAS is a 100 mm line with 'not alert' and 'alert' anchoring each end of the line. This is scored from mm distance along the line towards 'alert'; with a higher score indicating greater alertness.
Physical fatigue/ sleep quality | 56 days
  This outcome will be assessed via changes on the Athens Insomnia Scale (within the MFI-20). This is scored as per the MFI detailed in outcome 2 above.
Cognitive function | 56 days
  This outcome will be assessed via changes on the cognitive task outcomes (measured via COMPASS). COMPASS is a proprietorial software platform for delivering a range of cognitive tasks; assessing domains like memory and attention, with tasks scored for accuracy (% correct) and speed (msec).
Physiological induced stress | 56 days
  This outcome will be assessed via changes in heart rate (beats per minute) during the observed multitasking stressor. Higher values indicate greater stress.
Psychological induced stress | 56 days
  This outcome will be assessed via changes on the State portion Trait Anxiety Inventory (STAI). The state portion of this questionnaire comprises 20 items which is scored from 1 (not at all) to 4 (very much so) with a higher score indicating greater stress.
Galvanic skin response | 56 days
  This outcome will be assessed via changes in galvanic skin response (micro siemans) during the observed multitasking stressor). Higher values indicate greater stress.
Salivary cortisol | 56 days
  This outcome will be assessed via changes in salivary cortisol (nmol/L) during the observed multitasking stressor. Higher values indicate greater stress.
Alpha Amylase | 56 days
  This outcome will be assessed via changes in alpha amylase (nmol/L) during the observed multitasking stressor. Higher values indicate greater stress.

CONTACTS AND LOCATIONS:
Overall Officials: Emma Wightman, PhD, Principal Investigator — Northumbria University
Locations (1):
- Brain Performance and Nutrition Research Centre, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The is no plan to share the raw individual participant data with anyone other than the research team here at Northumbria University and the study sponsor.